CLINICAL TRIAL: NCT06171542
Title: Efficacy of a Single Image Guided Injection of Connective Tissue Matrix for Glenohumeral Arthritis
Brief Title: Efficacy of a Single Image Guided Injection of CTM for Glenohumeral Arthritis
Acronym: HC22-1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indiana Hand to Shoulder Center (Other)
Collaborators: CTM Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHTSC CTM Project HC22-2
Record Dates: First submitted 2023-12-01; First posted 2023-12-14 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis Shoulder; Glenohumeral Osteoarthritis; Shoulder Osteoarthritis

STUDY DESIGN:
Intervention Model Description: All glenohumeral joint injections will be performed by a physician under the guidance of either ultrasound or fluoroscopy to ensure and document intra-articular needle placement. 2cc of CTM Flow will be injected. The glenohumeral joint will be injected with the medication under the discretion of the treating surgeon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CTM Shoulder Injection (Experimental)
  Interventions: Device: CTM Injection

INTERVENTIONS:
Device: CTM Injection — All glenohumeral joint injections will be performed by a physician under the guidance of either ultrasound or fluoroscopy to ensure and document intra-articular needle placement. 2cc of CTM Flow will be injected. The glenohumeral joint will be injected with the medication under the discretion of the treating surgeon.

SUMMARY:
CTM Biomedical markets and distributes decellularized particulate human placental connective-tissue matrix products, intended solely for homologous use to supplement or replace damaged or inadequate connective-tissue. These are structural tissue allografts processed according to the criteria contained in 21CFR 1271.10(a) for regulation solely under section 361 of the Public Health Service Act.

The goal of this study is to determine the success rate of a single, image guided glenohumeral CTM injection (for radiographically confirmed glenohumeral osteoarthritis at follow up intervals of 1, 2, 3, 4, 6, 9, and 12 months. This will be measured using the Likert Pain Scale (LPS) and Oxford Shoulder Score (OSS). Secondary goals are to identify if certain demographic or imaging factors exist that predict early symptom recurrence requiring additional intervention, defined as a second connective tissue matrix injection, a subsequent corticosteroid injection, or arthroplasty.

DETAILED DESCRIPTION:
A recent prospective study by our center identified a clinically meaningful and statistical improvement after corticosteroid injection in the Oxford Shoulder Score and VAS pain scores in patients with glenohumeral arthritis2.

CTM Biomedical markets and distributes decellularized particulate human placental connective-tissue matrix products, intended solely for homologous use to supplement or replace damaged or inadequate connective-tissue. These are structural tissue allografts processed according to the criteria contained in 21CFR 1271.10(a) for regulation solely under section 361 of the Public Health Service Act. CTM Flow is decellularized particulate human placental connective-tissue matrix provided in a vial.

Osteoarthritis creates pain due to damaged tissues. CTM has been approved to supplement and replace damaged tissues. It is not replacing the damaged cartilage with new cartilage, but rather with other connective tissues. Previous unpublished studies in tonsil surgery and knee arthritis surgery have shown improvement from the CTM injections.

Image guided injection of the glenohumeral joint has been shown to be more accurate than blind in-office injections and will thus be used in this study3.

The goal of this study is to determine the success rate of a single, image guided glenohumeral (GH) CTM injection (for radiographically confirmed glenohumeral osteoarthritis at follow up intervals of 1, 2, 3, 4, 6, 9, and 12 months. This will be measured using the Likert Pain Scale (LPS) and Oxford Shoulder Score (OSS). Secondary goals are to identify if certain demographic or imaging factors exist that predict early symptom recurrence requiring additional intervention, defined as a second connective tissue matrix injection, a subsequent corticosteroid injection, or arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Radiographic documented Glenohumeral osteoarthritis (grade 1-3)
2. Males or females age 18 or older
3. Patients receiving a CTM injection for their initial treatment
4. Patients who can consent to be a part of this study
5. Patients who are able keep up regular communication through phone calls or electronic PROs

Exclusion Criteria:

1. Inflammatory Arthritis
2. Brachial Plexopathy
3. Cervical spine abnormalities such as radiculopathies
4. age less than 18 years
5. those unable to keep up monthly communication through phone calls and/or electronic PROs
6. Absence of glenohumeral osteoarthritis
7. Pregnancy or breastfeeding
8. Non-english speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Likert Pain Scale | 12 Months
  PROM
Oxford Shoulder Score | 12 Months
  PROM

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Hand to Shoulder Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No